CLINICAL TRIAL: NCT07018804
Title: Analysis of the Pathogenic Mechanism of Abnormal Airway Basal Cell Function in Bronchiolitis Obliterans Syndrome and Research on Targeted Treatment Strategies
Brief Title: Mechanisms and Targeted Therapy of Airway Basal Cell Dysfunction in Bronchiolitis Obliterans Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Haikou Affiliated Hospital of Central South University Xiangya School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SC20250160
Record Dates: First submitted 2025-05-17; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Bronchiolitis Obliterans Syndrome (BOS)
Keywords: Bronchiolitis Obliterans Syndrome; Airway epithelium; Airway basal cells; Inflammatory response
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Cloning, Organism; Gene Editing

STUDY DESIGN:
Intervention Model Description: In this experiment, bronchoscopic brushing was used to collect epithelial mucosal tissues from the diseased lung area and the relatively healthy lung lobe area of the patients. When conditions permit, alveolar lavage fluid specimens of the patients were collected simultaneously to isolate distal small airway stem cells. Allelic samples from healthy volunteers with no obvious airway abnormalities were used as parallel controls. The collected samples were digested with tissue collagenase and then used for the culture of airway BCS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Patient group (Experimental): Epithelial mucosal tissues from the diseased lung regions and relatively healthy lung lobes of BOS patients following hematopoietic stem cell transplantation (HSCT) will be collected. Alveolar lavage fluid specimens will be obtained when available. The intervention consists of digesting the collected samples with tissue collagenase for the culture of airway basal cells (BCs).
  Interventions: Procedure: Bronchoscopic brushing
- Healthy control group (Experimental): Healthy volunteers with no obvious airway abnormalities will be selected to collect samples from the same anatomical sites. No disease-related interventions will be performed, serving as a comparative control to highlight the abnormal conditions of basal cells (BCs) in the patient group.
  Interventions: Procedure: Bronchoscopic brushing
- Single - cell clone group (Experimental)
  Interventions: Genetic: Single - cell cloning
- Cell Function Identification Group (Experimental)
  Interventions: Genetic: Cell function identification
- Local microenvironment change identification group (Experimental)
  Interventions: Genetic: Identification of local microenvironmental changes
- Gene Editing Group (Experimental)
  Interventions: Genetic: Gene editing
- Ferret airway basal cell transplantation group (prevention group) (Experimental)
  Interventions: Procedure: Prevention of ferret airway basal cell transplantation
- Ferret airway basal cell transplantation group (treatment group) (Experimental)
  Interventions: Procedure: Transplantation treatment of ferret airway basal cells

INTERVENTIONS:
Procedure: Bronchoscopic brushing — The collected samples are digested with tissue collagenase for the culture of airway basal cells (BCs).
  Arms: Healthy control group; Patient group
Genetic: Single - cell cloning — After primary BCs are expanded in the P1 passage, single-cell cloning libraries are established by planting them into 384-well cell culture plates in a single-cell per well format using a flow chamber cell sorter. Ten samples are selected from the expandable clones for the identification of differentiation and proliferation capabilities, while the remaining clones are cryopreserved.
  Arms: Single - cell clone group
Genetic: Cell function identification — For single-cell samples of each patient, in vitro expansion culture is performed to observe the morphology of cells at each passage and calculate the clonogenic rate. Immunofluorescence technique is used to detect the expression of the cell proliferation marker Ki67, and the proliferation capacity is evaluated by combining with the CCK8 assay. Cells at passages P3-P5 are seeded on the permeable membrane of cell culture inserts at a density of \(10^6\) cells/cm², and after 21 days of culture, the differentiated structures are collected. The expression of ciliated cell marker Ace-Tubulin and goblet cell marker MUC5AC is detected to assess the differentiation capacity. Meanwhile, cells are injected subcutaneously into NSG mice at \(10^6\) cells/injection site for in vivo differentiation for 28 days, and the differentiated structures are collected for pathological analysis.
  Arms: Cell Function Identification Group
Genetic: Identification of local microenvironmental changes — The air-liquid interface (ALI) differentiation culture medium is collected, and cell debris is removed by high-speed centrifugation. The supernatant is then collected to extract proteins. Target proteins are purified via immunoprecipitation or affinity chromatography, followed by desalting and concentration for mass spectrometry analysis to detect inflammatory cytokines and extracellular matrix (ECM). Real-time PCR and Western blot techniques are used to measure the expression levels of epithelial markers, mesenchymal markers, and ECM in cells across all groups, thereby evaluating changes in the local microenvironment around small airways.
  Arms: Local microenvironment change identification group
Genetic: Gene editing — After plasmid construction, based on gene function, the CRISPR-Cas9-sgRNA (all-in-one) plasmid is transiently transfected into expanded single-cell strains via Nucleofection to knockout the target gene, or the CRISPR-dCas9 fusion-sgRNA plasmid is transiently transfected to activate or inhibit the target gene. After 3-5 days of culture, viable cells are sorted by FACS, and single cells are seeded into 96-well plates for two additional passages of expansion. Samples are collected for Sanger sequencing to screen successfully constructed cell lines.
  Arms: Gene Editing Group
Procedure: Prevention of ferret airway basal cell transplantation — Before surgery, basal cells (BCs) of recipient ferrets are collected by bronchoscopic brushing, followed by in vitro culture and identification. Prior to the onset of BOS, the cells are injected into recipient ferrets via bronchoscopy. Outcomes including ferret survival rate, body weight, CT imaging, and lung tissue pathology are collected to evaluate the preventive effect of BCs on BOS.
  Arms: Ferret airway basal cell transplantation group (prevention group)
Procedure: Transplantation treatment of ferret airway basal cells — Stable cell lines with target gene knockdown are established in ferret basal cells (BCs). After ferrets develop bronchiolitis obliterans syndrome (BOS), the constructed cell lines are transplanted into recipient ferrets to validate the therapeutic effect of gene-corrected BCs on the disease.
  Arms: Ferret airway basal cell transplantation group (treatment group)

SUMMARY:
This experimental study aims to investigate the pathogenesis of bronchiolitis obliterans syndrome (BOS) and provide a basis for clinical diagnosis and treatment. The core research question is: whether there is a causal relationship between stem cell dysfunction induced by the inflammatory microenvironment and airway injury repair during the pathological process of BOS? Researchers will collect alveolar lavage fluid specimens from participants and healthy individuals to isolate distal small airway stem cells for subsequent scientific research and comparative analysis, thereby revealing the pathological mechanisms of BOS, exploring precise intervention targets, and developing innovative therapeutic strategies to improve patient prognosis, long-term survival rates, and quality of life.

DETAILED DESCRIPTION:
The purpose of this experimental study is to explore the role of airway basal cells in the development of bronchiolitis obliterans syndrome (BOS) and develop potential therapeutic strategies. The main question it aims to answer is: How do the functional abnormalities of airway basal cells (BCs) affect the progression of BOS and what are the underlying molecular mechanisms? Researchers will collect epithelial mucosal tissues from diseased and relatively healthy lung regions of BOS patients through bronchoscopic brushing, and simultaneously gather alveolar lavage fluid specimens when possible. Specimens from healthy volunteers with no obvious airway abnormalities will be used as controls. After that, BCs will be isolated from these specimens. The isolated BCs will be cultured and their molecular characteristics will be identified using immunofluorescence staining to detect the expression of BCs markers such as p63 and Krt5.

Subsequently, single - cell clone libraries will be established by flow cytometry cell fluorescence sorting (FACS) technology. Multiple aspects of the cells' functions will be evaluated, including self - renewal ability by detecting the expression of the proliferation marker Ki67 through immunofluorescence and CCK8 assay, and differentiation ability by analyzing the cell types and proportions in the differentiation structures of in vitro air - liquid interface (ALI) culture for 21 days and in vivo differentiation in severe combined immunodeficiency (NSG) mice for 28 days using Real - time PCR and immunofluorescence techniques.

In addition, multi - omics sequencing technologies, such as RNA - seq, ATAC - seq, and CUT&Tag, will be employed to explore the molecular mechanisms of BCs' functional abnormalities. Stable interference cell lines will be established using CRISPR - Cas9 technology to verify the functions of potential target genes. A ferret BOS model will be constructed, and BCs transplantation experiments will be carried out in ferrets. By observing and analyzing the survival rate, body weight, CT images, and lung tissue pathology of ferrets, the preventive and therapeutic effects of BCs on BOS will be evaluated.

By clarifying the role of BCs in BOS, this study aims to reveal the underlying pathological mechanisms, explore potential intervention targets, and develop novel treatment approaches. These efforts are expected to improve the prognosis of BOS patients, reduce the incidence and mortality rates, and enhance the overall quality of life for those affected by this life - threatening respiratory disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received allogeneic hematopoietic stem cell transplantation and are diagnosed with bronchiolitis obliterans syndrome

Exclusion Criteria:

* Bronchoscopy consultation is not suitable for patients who are not suitable for bronchoscopy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The self - renewal ability of airway basal cells | From enrollment to 32 weeks
  By comparing the Ki67 expression levels of airway basal cells and the results of the CCK8 assay in different samples (such as patients with bronchiolitis obliterans syndrome and healthy volunteers), clarify the abnormal manifestations of the self - renewal function of airway basal cells in the disease state, and further explore the internal connection between it and the occurrence and development of bronchiolitis obliterans syndrome.
Differentiation ability of airway basal cells | From enrollment to 32 weeks
  Collect the differentiation samples of the air - liquid interface (ALI) in vitro differentiation culture for 21 days and the severe combined immunodeficiency (NSG) mice in vivo differentiation for 28 days respectively. With the help of real - time fluorescence quantitative polymerase chain reaction (Real - time PCR) and immunofluorescence techniques, conduct a detailed analysis of the cell types and their proportions in the differentiated structures. By detecting the expression of ciliated cell marker Ace - Tubulin, goblet cell marker MUC5AC, etc., accurately evaluate the ability of airway basal cells to differentiate into different cell types, providing a key basis for a deep understanding of the mechanism of airway epithelial injury repair.
Survival rate of ferret experiments | From enrollment to 32 weeks
  In the ferret airway basal cell transplantation experiment, closely monitor the survival rate of ferrets, which is a key indicator for evaluating the impact of airway basal cell transplantation on the disease progression of bronchiolitis obliterans syndrome.
Weight changes in ferret experiments | From enrollment to 32 weeks
  In the experiment of ferret airway basal cell transplantation, the weight changes of ferrets are regularly recorded. The weight changes can intuitively reflect the overall health of ferrets and assist in judging the effect of airway basal cell transplantation.

SECONDARY OUTCOMES:
Molecular characteristics of cells | From enrollment to 32 weeks
  The immunofluorescence staining experiment was used to observe the expression of airway basal cell markers, such as transformation protein 63 (p63) and keratin 5 (Krt5). By detecting the expression of these markers, it was possible to accurately determine whether the cultured cells were airway basal cells, providing a reliable guarantee of cell sources for subsequent experiments.
Microenvironment change | From enrollment to 32 weeks
  Collect the gas - liquid interface (ALI) differentiation medium, remove cell debris by high - speed centrifugation, and collect the supernatant. Extract the proteins in the supernatant, purify the target protein using immunoprecipitation or affinity chromatography techniques. After desalting and concentration, perform mass spectrometry analysis, and quantitatively detect inflammatory cytokines and extracellular matrix. At the same time, use real - time fluorescence quantitative polymerase chain reaction (Real - time PCR) and Western blot techniques to detect the expression levels of epithelial markers, mesenchymal markers, and extracellular matrix in cells of each group, comprehensively evaluate the changes in the local microenvironment around the small airways, and reveal the interaction mechanism between the microenvironment and the function of airway basal cells.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Yang, DM, Principal Investigator — Department of Hematology, Haikou People's Hospital
Locations (1):
- Haikou Affiliated Hospital of Central South University Xiangya School of Medicine, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No
The IPD encompasses highly sensitive and confidential data that was collected through significant investment of our resources, both in terms of time and funding. This data is integral to our ongoing research initiatives, which are at a crucial stage of development. Premature sharing could disrupt our research timelines and strategic plans. Additionally, we have not yet established comprehensive safeguards to ensure that the data will be used appropriately by external researchers. Without proper protocols in place, there is a risk of misuse or misinterpretation of the data, which could lead to inaccurate research outcomes and potential reputational damage to our institution. For these reasons, we have decided not to share the IPD at this time.